CLINICAL TRIAL: NCT06371547
Title: Efficiency of Different Types of Stretching Exercises on Gastrocnemius Tightness
Brief Title: Efficiency of Different Gastrocnemius Stretching Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEUFTR-3
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-12

CONDITIONS: Muscle Tightness
Keywords: pain threshold; elasticity
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Interventions and assessment will be performed by separate researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sustained stretching of the gastrocnemius muscle with a towel (Experimental): The participant will place a towel under the plantar surface of the foot and, using both hands, pull the towel towards themselves until they feel a stretch in the calf muscle. Subsequently, they will be asked to maintain this position for 3 minutes. The stretching exercise will be performed in 3 sets per day.
  Interventions: Other: Stretching Exercise
- Intermittent stretching of the gastrocnemius muscle with a towel (Experimental): In intermittent stretching with a towel, the individual will place a towel under the plantar surface of the foot and, using both hands, pull the towel towards themselves until they feel a stretch in the calf muscle. Subsequently, they will be instructed to maintain this position for 20 seconds. The stretching exercise will be performed in 2 sets per day, with 5 repetitions in each set.
  Interventions: Other: Stretching Exercise
- Sustained stretching against the wall (Experimental): In sustained stretching against the wall, individuals will be asked to place their hands on the wall at shoulder width apart. One leg will be positioned behind the other. Then, the front knee will be bent while keeping the back knee in extension and the heel in contact with the ground. Individuals will be instructed to bend their knees until they feel a stretch in the calf muscle. Subsequently, they will be asked to maintain this position for 3 minutes. The stretching exercise will be performed in 3 sets per day.
  Interventions: Other: Stretching Exercise
- Intermittent stretching against the wall (Experimental): During intermittent stretching against the wall, individuals will be instructed to place their hands on the wall at shoulder width apart. One leg will be positioned behind the other. Then, the knee of the front leg will be bent while the knee of the back leg continues to stay in extension, and the heel remains in contact with the ground. Individuals will be asked to bend their knee until they feel a stretch in the calf muscle. Subsequently, they will be instructed to maintain this position for 20 seconds. The stretching exercise will be performed in 2 sets per day, with 5 repetitions in each set.
  Interventions: Other: Stretching Exercise

INTERVENTIONS:
Other: Stretching Exercise — Participants will perform different types and durations of gastrocnemius muscle stretching exercises according to their assigned groups for two weeks.

SUMMARY:
The primary aim of this study is to investigate the effects of different types and durations of gastrocnemius stretching on the viscoelastic properties of the gastrocnemius muscle, Achilles tendon, and plantar fascia.In addition, pain threshold of the gastrocnemius muscle and plantar fascia, as well as on hamstring tightness will be measured.

DETAILED DESCRIPTION:
The study will include a total of at least 48 individuals who meet the inclusion and exclusion criteria. Subsequently, participants will be randomly assigned to one of four groups for gastrocnemius stretching exercises of different durations and types. Participants in Group I will perform sustained stretching with a towel, those in Group II will perform intermittent stretching with a towel, those in Group III will perform sustained stretching against the wall, and those in Group IV will perform intermittent stretching against the wall. The stretching exercises will be performed under the supervision of one of the researcher. Compliance with the stretching exercise will be evaluated by keeping a daily log.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 25 years
* Having a gastrocnemius muscle tightness in the dominant side

Exclusion Criteria:

* History of lower extremity surgery or trauma
* Diagnosis of fibromyalgia, neurological disease, achilles tendinopathy, metatarsalgia, acute ankle sprain, tarsal tunnel syndrome, or heel pad syndrome
* Having received physiotherapy related to the lower extremities within the last six months
* A body mass index (BMI) above 30 kg/m2
* Having received a local steroid injection within the last six weeks
* The presence of a local infection
* The presence of rheumatic or other systemic inflammatory diseases
* Diabetes or other metabolic diseases
* Nerve compression syndrome
* Currently using painkillers
* Diagnosis of neurological heel pain
* A positive navicular drop test result
* Having engaged in strenuous exercise within the last 24 hours
* Not being fully compliant with the exercise program

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of the Viscoelastic Properties | Change from baseline viscoelastic properties at seventh and fourteen day
  The effect of stretches on the viscoelastic properties of the stretched muscle and its associated anatomical regions will be evaluated non-invasively using the myotonometer. Measurements will be taken on the medial and lateral gastrocnemius, Achilles tendon, and plantar fascia. The measurement areas will be marked prior to measurement. Measurements of the gastrocnemius and Achilles tendon will be taken with individuals lying prone, knees extended, and ankles in a neutral position. Measurement of plantar fascia tone will be taken with individuals lying prone, hips in neutral, knees extended, ankles in neutral position with goniometer assistance, and supported. All measurements will be taken three times, and the averages will be recorded.
Ankle-foot Dorsiflexion Index | Change from baseline ankle dorsiflexion range of motion at seventh and fourteen day
  The ankle-foot dorsiflexion index will be used to assess both the tightness of the gastrocnemius muscle and the effectiveness of stretches. The individual's dorsiflexion range of motion will be measured using the lunge test, with measurements taken in both knee extension and flexion positions, and the difference between these measurements will be recorded as the ankle-foot dorsiflexion index.

SECONDARY OUTCOMES:
Measurement of the Mechanosensitivity | Change from baseline pain at seventh and fourteen day
  The effect of stretching on pain threshold will be assessed using an analog algometer. Pain threshold measurements will be taken on the gastrocnemius and plantar fascia. The measurement points for the gastrocnemius muscle will be the same as the viscoelastic measurement points. The measurement point for the plantar fascia will be the point where the plantar fascia attaches to the heel. Pain threshold measurements will be taken with the individual lying prone, with their feet hanging off the treatment bed. Measurements will be taken at each point with a 30-second interval, and three measurements will be taken for each point. The averages of these measurements will be calculated.
Assessment of Hamstring Tightness | Change from baseline hamstring tightness at seventh and fourteen day
  The hamstring muscle tightness in the individuals participating in the study will be assessed using the straight leg raise test. The straight leg raise test is particularly used to evaluate the tightness and elasticity of the hamstring muscles. For the test, the individual will be positioned in a supine lying position with the hip and knee joints in a neutral position. Subsequently, while the knee is in extension, the hip will gradually be brought into flexion. Hip flexion will be stopped when the individual feels discomfort from the tension behind the hip. Then, using a goniometer, the angle formed between the individual's lower extremity and the treatment bed will be measured. The center of the goniometer will be placed on the greater trochanter, with one arm along the lateral thigh and the other arm parallel to the treatment bed. An angle of 80 degrees is considered normal. The measurement will be repeated three times, and the average of the three measurements will be calculated.

OTHER OUTCOMES:
Dominant Leg Determination | At the baseline
  To determine the dominant lower extremity of the individuals to be included in the study, they will be asked the question 'which foot do you use to kick a ball?
Navicular Drop Test | At the baseline
  The navicular drop test will be used to evaluate the medial longitudinal arch of the individuals participating in the study. The test will be performed in two different positions: sitting and standing. First, in the sitting position, the navicular tuberosity of the individual will be marked with a pen, and the distance to the ground will be measured. Then, the individual will be asked to stand up and transfer all body weight onto their feet, and again the distance between the navicular tuberosity and the ground will be measured. A difference of more than 10 mm between the two measurements indicates that the individual's foot is in pronation.
Self-reported Effects of Stretching Exercises | Change from baseline self-reported effects of stretching exercises at seventh and fourteen day
  "Participants in the study will be asked to mark any symptoms such as muscle fatigue or pain they experience in any part of their body on a body diagram and rate the severity of these symptoms on a numeric rating scale from 0 to 10."
The Satisfaction Level with the Stretching | Change from baseline at seventh and fourteen day
  The satisfaction level with the stretching treatment will be evaluated using the Numeric Rating Scale (NRS). Participants will be asked to rate their satisfaction level with the stretching treatment, and they will be asked to score between 0% and 100%. A score of 0% indicates 'no effect' while 100% indicates 'very satisfied'.
Compliance with Stretching Exercise Program | Change from baseline at fourteen day
  The participants' compliance with the stretching exercise program was categorized based on the percentage of required sets and repetitions completed: (1) fully compliant if 85% were completed, (2) partially compliant if 70% to 84% were completed, (3) poorly compliant if 50% to 69% were completed, and (4) noncompliant if 10% to 49% were completed.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; Erhan Dincer, M.Sc., Principal Investigator — Bitlis Eren University; Cihan Önen, Asst. Prof., Principal Investigator — Bitlis Eren University; Abdurrahman Tanhan, Ph.D., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cullen NP, Singh D. Plantar fasciitis: a review. Br J Hosp Med (Lond). 2006 Feb;67(2):72-6. doi: 10.12968/hmed.2006.67.2.20465. No abstract available. PMID 16498906
- [Background] Schwartz EN, Su J. Plantar fasciitis: a concise review. Perm J. 2014 Winter;18(1):e105-7. doi: 10.7812/TPP/13-113. PMID 24626080
- [Background] Porter D, Barrill E, Oneacre K, May BD. The effects of duration and frequency of Achilles tendon stretching on dorsiflexion and outcome in painful heel syndrome: a randomized, blinded, control study. Foot Ankle Int. 2002 Jul;23(7):619-24. doi: 10.1177/107110070202300706. PMID 12146772
- [Background] Liu CL, Li YP, Wang XQ, Zhang ZJ. Quantifying the Stiffness of Achilles Tendon: Intra- and Inter-Operator Reliability and the Effect of Ankle Joint Motion. Med Sci Monit. 2018 Jul 14;24:4876-4881. doi: 10.12659/MSM.909531. PMID 30006997
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Weerasinghe TW, Goonetilleke RS, Reischl U. Pressure thresholds and stiffness on the plantar surface of the human foot. Ergonomics. 2017 Jul;60(7):985-996. doi: 10.1080/00140139.2016.1229042. Epub 2016 Sep 26. PMID 27609429
- [Background] Ajimsha MS, Binsu D, Chithra S. Effectiveness of myofascial release in the management of plantar heel pain: a randomized controlled trial. Foot (Edinb). 2014 Jun;24(2):66-71. doi: 10.1016/j.foot.2014.03.005. Epub 2014 Mar 21. PMID 24703512
- [Background] Bolivar YA, Munuera PV, Padillo JP. Relationship between tightness of the posterior muscles of the lower limb and plantar fasciitis. Foot Ankle Int. 2013 Jan;34(1):42-8. doi: 10.1177/1071100712459173. PMID 23386760
- [Background] McPoil TG, Cornwall MW. The relationship between static lower extremity measurements and rearfoot motion during walking. J Orthop Sports Phys Ther. 1996 Nov;24(5):309-14. doi: 10.2519/jospt.1996.24.5.309. PMID 8902683
- [Background] Naruseviciute D, Kubilius R. The effect of high-intensity versus low-level laser therapy in the management of plantar fasciitis: randomized participant blind controlled trial. Clin Rehabil. 2020 Aug;34(8):1072-1082. doi: 10.1177/0269215520929073. Epub 2020 Jun 8. PMID 32513018
- [Background] Monteagudo M, de Albornoz PM, Gutierrez B, Tabuenca J, Alvarez I. Plantar fasciopathy: A current concepts review. EFORT Open Rev. 2018 Aug 29;3(8):485-493. doi: 10.1302/2058-5241.3.170080. eCollection 2018 Aug. PMID 30237906
- [Background] Hirata K, Kanehisa H, Miyamoto N. Acute effect of static stretching on passive stiffness of the human gastrocnemius fascicle measured by ultrasound shear wave elastography. Eur J Appl Physiol. 2017 Mar;117(3):493-499. doi: 10.1007/s00421-017-3550-z. Epub 2017 Feb 4. PMID 28161870
- [Background] Kanehisa H, Ikegawa S, Tsunoda N, Fukunaga T. Cross-sectional areas of fat and muscle in limbs during growth and middle age. Int J Sports Med. 1994 Oct;15(7):420-5. doi: 10.1055/s-2007-1021081. PMID 8002122
- [Background] Masood T, Bojsen-Moller J, Kalliokoski KK, Kirjavainen A, Aarimaa V, Peter Magnusson S, Finni T. Differential contributions of ankle plantarflexors during submaximal isometric muscle action: a PET and EMG study. J Electromyogr Kinesiol. 2014 Jun;24(3):367-74. doi: 10.1016/j.jelekin.2014.03.002. Epub 2014 Mar 20. PMID 24717406
- [Background] Kamonseki DH, Goncalves GA, Yi LC, Junior IL. Effect of stretching with and without muscle strengthening exercises for the foot and hip in patients with plantar fasciitis: A randomized controlled single-blind clinical trial. Man Ther. 2016 Jun;23:76-82. doi: 10.1016/j.math.2015.10.006. Epub 2015 Oct 30. PMID 26654252